CLINICAL TRIAL: NCT07193550
Title: A Phase 2 Trial of Zanzalintinib in Advanced/Metastatic Bone Sarcomas (ZAMBONE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0912
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bone Sarcomas
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 2 Cohorts A, B, C, D: Treatment with Zanzalintinib (Experimental): Four cohorts of patients based on biology of the disease will be included in this trial:
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — Participants will take zanzalintinib 100mg daily by mouth
  Other Names: XL092

SUMMARY:
To study the treatment efficacy of zanzalintinib monotherapy in patients with advanced and/or metastatic bone sarcomas.

DETAILED DESCRIPTION:
Primary Objectives:

* For cohort A (osteosarcoma) progression-free survival (PFS) rate at 16 weeks (PFS16 weeks)
* For cohort B (Ewing sarcoma), cohort C (chondrosarcoma), and cohort D (other bone sarcomas), progression-free survival (PFS) at 12 weeks (PFS12 weeks).

Secondary Objectives:

* To estimate the objective response rate (ORR) within each cohort by RECIST 1.1 criteria.
* To estimate the progression-free survival (PFS) and overall survival in patients with locally advanced or metastatic bone sarcomas receiving zanzalintinib.
* To evaluate the safety and tolerability of zanzalintinib within each cohort and across cohorts as assessed by toxicity rates according to CTCAE version 5.0 criteria.

Exploratory Objectives:

To determine the expression of selected biomarkers in pre-treatment and on-treatment tumor biopsy specimens and correlate with clinical benefit within each cohort and across cohorts

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥ 18 years old with pathologically confirmed unresectable locally advanced or metastatic bone sarcoma in one of the following categories: Cohort A - Osteosarcoma, Cohort B - Ewing sarcoma, Cohort C - Chondrosarcoma (conventional, grades 2-3), Cohort D - Other primary sarcoma of bone including but not limited to dedifferentiated chondrosarcoma, undifferentiated pleomorphic sarcoma (UPS) of bone, chordoma, and non-Ewing's round cell sarcomas of bone.

chondrosarcoma, undifferentiated pleomorphic sarcoma (UPS) of bone, chordoma, and non-Ewing's round cell sarcomas of bone.

* Patients with conventional chondrosarcoma (Cohort C) must demonstrate evidence of disease progression by RECIST 1.1 within 12 weeks of trial enrollment

  * Patients must have relapsed or become refractory to conventional therapy, receiving at least 1 prior line of systemic therapy unless no standard of care exists.
  * Patients may have received no more than 2 prior lines of systemic therapy in the advanced/metastatic setting.
* Multi-agent and/or alternating neoadjuvant/adjuvant standard of care chemotherapy will be counted as 1 line of systemic therapy if given for metastatic disease. Otherwise, neoadjuvant/adjuvant chemotherapy for localized disease does not apply towards the limitation regarding prior lines of systemic therapy.

  * Patients must have a performance status corresponding to ECOG scores of 0, 1 or 2 (Karnofsky ≥60%).
  * Weight >/= 40 kg.
  * Patients must have measurable disease per RECIST v1.1
  * Prior radiation will be allowed assuming there is measurable disease based upon RECIST 1.1 and at least 21 days from the completion of all radiation prior to initiation of study treatment. (Note: Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation)
  * Hematological function, as follows:
* Absolute neutrophil count (ANC) ≥ 1500/mm3 (growth factor/G-CSF permitted)
* Platelet count ≥ 100,000/mm3
* Hemoglobin > 9 g/dL.

  * INR ≤ 1.5 and activated partial thromboplastin time (aPTT) < 1.2 x upper limit of normal (ULN), except subjects on anticoagulation.
  * Renal function as follows: calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft Gault equation.
  * Hepatic function as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN and total bilirubin ≤ 1.5 x ULN (for subjects with Gilberts's disease ≤ 3 x ULN), serum albumin ≥ 2.
  * All patients must agree to consent and co-enroll on MD Anderson MOSAIC protocol to allow for sample collection and correlative studies
  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
  * Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
  * Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
  * Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
  * Sexually active fertile subjects and their partners must agree to use highly effective method of contraception (hormonal or barrier method of birth control, intrauterine device, tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, condoms, or abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

In addition, men must agree not to donate sperm through 96 days after the last dose of zanzalintinib and women (WOCBP) must agree not to donate effs (ova, oocyte) for the purpose of reproduction for at least 186 days after the last dose of zanalintinib.

• Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Prior treatment with zanzalintinib.

* Patients with primary soft tissue sarcoma with metastasis to bone.

  o Patients with histologically confirmed Ewing's sarcoma with either bone or soft tissue primary site are eligible for enrollment in Cohort B
* Patients with known sensitivity to the study agents and/or previously identified allergy or hypersensitivity to components of treatment
* Patients previously treated with other VEGF-targeted TKIs (including but not limited to cabozantinib, regorafenib, pazopanib, or similar).
* Receipt of any small molecule kinase inhibitor (including investigational within 2 weeks before first dose of study treatment.
* Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression.
* Active infection requiring intravenous (IV) antibiotics within 2 weeks of study enrollment.
* Prior receipt of an investigational study drug and/or procedure within 21 days of study day 1.
* Anti-tumor therapy within 21 days of study day 1 including chemotherapy, antibody therapy, or other investigational agent.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks, or systemic treatment with radionuclides within 6 weeks before first dose of study treatment; ongoing clinically relevant complications from prior radiation therapy are not eligible.
* Any complementary medicine such as herbal supplements, Chinese medicines, or other non-prescription medications being used for the treatment of bone sarcoma within 2 weeks prior to first dose of treatment as detailed in section5.5.
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class > II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry.
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C.
* Patients with known human immunodeficiency virus (HIV) infection with detectable viral load.

HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

* Known infection with acute or chronic hepatitis B or C.
* History of solid organ or allogeneic stem cell transplant
* Any other known concurrent or prior malignancy at time of or within 2 years of first does of study treatment. Prior malignancy that is in remission or otherwsie has not required treatment in > 2 years will be permitted.
* Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.
* Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment. Note, patients with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion) for at least 1 week before first dose of study treatment.
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  * Tumors invading the GI-tract from external viscera
  * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
  * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and asymptomatic
  * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months of the first dose. Note, complete healing of an intra-abdomninal abscess must be confirmed before first dose of study treatment
  * Known gastric or esophageal varices
  * Ascites, pleural effusion, or pericardial effusion requiring drainage in last 4 weeks
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Symptomatic cavitating pulmonary lesion(s) or endobronchial disease. Note, asymptomatic or radiated lesions allowed
* Lesions invading major blood vessel including but not limited to inferior vena cava, pulmonary artery, or aorta. Note, patients with intravascular tumor extension (i.e. tumor thrombus in renal vein or inferior vena cava) may be eligible following Principal Investigator approval
* Other clinically significant disorders that would preclude safe study participation:

  * Serious non-healing wound, ulcer, or bone fracture. Note, non-healing wounds or ulcers may be permitted if due to tumor associated skin lesions
  * Malabsoprtion syndromes
  * Pharmacologically uncompensated, symptomatic hypothyroidism
  * Requirement for hemodialysis or peritoneal dialysis
  * History of solid organ or allogeneic stem cell transplant
* Major surgery (i.e. GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laproscopic surgeries withint 4 weeks prior to first dose of study treatment. Minor surgery (i.e. simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment. Note, fresh/pre-treatment tumor biopsies should be completed at least 5 days prior to the first dose of study treatment. Patients with clinically relevant ongoing complications of prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 470 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment. Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because zanzalintinib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with zanzalintinib, breastfeeding should be discontinued if the mother is treated with zanzalintinib. These potential risks may also apply to other agents used in this study.
* Inability to swallow tablets or ingest a suspension either orally or by nasogastric (NG) or gastronomy (PEG) tube.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors ) and platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
  * Note, Subjects must have discontinued prohibited oral anticoagulants at least 3 days or 5 half-lives prior to the first dose of study treatment, whichever is longer
* Proteinuria > 1g/day.
* Other conditions, which in the opinion of the investigator, would compromise the safety of the patient's ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: John Livingston, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org